CLINICAL TRIAL: NCT06644339
Title: Remote Multichannel Monitoring of Patients With Chronic DIseAses Using Speech technoLogies Based On Artificial intelliGence
Acronym: DIALOG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Collaborators: PJSC VimpelCom (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIALOG2024
Record Dates: First submitted 2024-10-03; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Diabetes Mellitus; Arterial Hypertension; Lymphoproliferative Disease; Total Knee Replacement
Keywords: heart failure; diabetes mellitus; arterial hypertension; lymphoproliferative diseases; knee replacement; remote monitoring; mHealth; telemedicine; voice assistant
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus; Hypertension; Lymphoproliferative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Heart Failure (Experimental): Patients with chronic heart failure who was hospitalized due to decompensation of their condition. Their condition should be stabilized before discharge.
  Robotic remote monitoring of patients using unique algorithms developed for virtual operator speech technology and a BI system by voice commands to automate data collection and obtain information about the patient's well-being and his vital signs (blood pressure, heart rate, weight) related to heart failure.
  Interventions: Device: Voice assistant
- Diabetes mellitus (Experimental): Patients with diabetes mellitus who was hospitalized with unstable glucose level. Their condition should be stabilized before discharge.
  Robotic remote monitoring of patients using unique algorithms developed for virtual operator speech technology and a BI system by voice commands to automate data collection and obtain information about the patient's well-being and his vital signs (blood pressure, heart rate, weight, glucose) related to diabetes mellitus.
  Interventions: Device: Voice assistant
- Arterial hypertension (Experimental): Patients with arterial hypertension who was hospitalized with unstable arterial pressure. Their condition should be stabilized before discharge.
  Robotic remote monitoring of patients using unique algorithms developed for virtual operator speech technology and a BI system by voice commands to automate data collection and obtain information about the patient's well-being and his vital signs (blood pressure, heart rate, hypotension sings, signs of damage to target organs).
  Interventions: Device: Voice assistant
- Lymphoproliferative diseases (Experimental): Patients with any lymphoproliferative disease who is undergoing chemotherapy. Their condition should be stabilized before discharge.
  Robotic remote monitoring of patients using unique algorithms developed for virtual operator speech technology and a BI system by voice commands to automate data collection and obtain information about the patient's well-being and his vital signs (blood pressure, heart rate) related to chemotherapy complications.
  Interventions: Device: Voice assistant
- Total knee replacement (Experimental): Patients who underwent total knee replacement. Their condition should be stabilized before discharge.
  Robotic remote monitoring of patients using unique algorithms developed for virtual operator speech technology and a BI system by voice commands to automate data collection and obtain information about the patient's well-being and his vital signs (pain, fever) related to replacement complications.
  Interventions: Device: Voice assistant

INTERVENTIONS:
Device: Voice assistant — Robotic remote monitoring of patients using unique algorithms developed for virtual operator speech technology and a BI system by voice commands on the "question-answer" principle. It allows us to automate data collection and obtain information about the patient's well-being and his vital signs (blood pressure, heart rate, weight) depending on disease.
  Follow-up and management of disease provided by specialists at participating institutions.

SUMMARY:
DIALOG is a study to assess the efficacy and safety of remote patient monitoring using virtual operator voice technologies and a business intelligence (BI) system for timely detection, prevention of early complications, worsening of the condition, and other adverse events in patients who have been discharged from the hospital.

DETAILED DESCRIPTION:
After ensuring that the patient's characteristics meet the inclusion and exclusion criteria and confirming the patient's ability to use the "voice assistant", as provided in the research protocol, patients who have completed the briefing will be able to use the voice assistant at home. During the month, robotic remote monitoring of patients using unique algorithms developed for virtual operator speech technology and a BI system will be conducted for five groups of patients (CHF, DM, AH, LPD, and patients who underwent total knee replacement) who have been discharged from the hospital. The system developed allows for quick surveys, collection of data on patient conditions, and convenient transfer of this data to the physician. The physician will receive information on patient status in a graphical form using a traffic light system. In the event of any red flags, the physician will contact the patient for further discussion on treatment strategies. The study will evaluate the efficacy and safety of utilizing the "voice assistant" by assessing the achievement of target values for controlled parameters, evaluating patient satisfaction and adherence to treatment, reducing the number of repeat hospitalization, and reducing overall mortality and cardiovascular-related mortality.

ELIGIBILITY:
Inclusion Criteria:

* Disease diagnosed according to the latest Clinical practice guidelines
* Stable condition at the time of discharge from the hospital
* Written informed consent to participate in the study

Non-inclusion criteria:

* Diagnosed dementia or severe cognitive impairment
* The inability to use automatic devices to register blood pressure at home, a blood glucose meter
* Alcohol or drug abuse
* Inability to contact a voice assistant and other study requirements, due to major co-morbidities, social or financial issues, or a history of noncompliance with medical regimens, that might compromise the patient's ability to understand and/or comply with the protocol instructions or follow-up procedures

Exclusion Criteria:

* Unwillingness of the patient to continue participating in the study
* The development of conditions related to the criteria of non-inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
cardiovascular mortality | an average, 1 month after randomization
  mortality rate
all-cause mortality | an average, 1 months after randomization
  mortality rate
complications, decompensations | an average, 1 month after randomization
  rate of complications and exacerbations of the main disease

SECONDARY OUTCOMES:
achievement target or maximally tolerated doses | an average, 1 month after randomization
  achievement target or maximally tolerated doses for CHF, DM and AH
satisfaction | an average, 1 month after randomization
  satisfaction of patients and doctors with the robotic speech questionnaire
changes in medical adherence | an average, 1 month after randomization
  change in amount of taking drugs and doses

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kozhevnikova, Professor, Principal Investigator — The Sechenov First Moscow State Medical University
Locations (1):
- Federal State Autonomous Educational Institution of Higher Education I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University), University Clinical Hospital No.1, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
According to the Local Ethics Committee's rules, we are not allowed to provide this data.